CLINICAL TRIAL: NCT03939377
Title: Evaluation of an Osteopathic Procedure in the Management of Pain in Palliative Care Patients in a Mobile Palliative Care Support Team (EMASP): Controlled, Randomized, Single-blind Study
Brief Title: Osteopathic Procedure on Pain in Palliative Care
Acronym: OSTEOPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OSTEOPAL; 2018-A02655-50 (Other: ID-RCB)
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Pain
Keywords: Palliative; Osteopathy
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathy (Experimental): Management will be centered on the skull, the sacrum, the cranio-sacral axis, the entire visceral abdominal and thoracic system.
  Interventions: Other: Questionnaire and treatment
- Simulate (Placebo Comparator): The simulated treatment will be characterized by placing the practitioner's hands on the patient in the areas tested without any intention of treatment.
  Interventions: Other: Questionnaire and treatment

INTERVENTIONS:
Other: Questionnaire and treatment — EVA questionnaire every day for 7 days. treatment (real or simulated) at J3 and J5

SUMMARY:
The culture of the palliative is anchored more and more in France. In 2009, nearly 9 out of 10 French people (89%) believe that palliative care can reduce the suffering of people at the end of their lives. Despite the rise of palliative care in France, their access is not homogeneous between regions. In 2010, it is estimated that 2 French out of 3 likely to receive palliative care could not access it. Palliative care remains essential at the end of the patient's life, as well as for the family and caregivers.

The French government has put in place three national palliative care development programs: 2002-2005, 2008-2012, 2015-2018. The last program has unlocked a budget of 190 million euros for their development. It has been estimated from Social Security reimbursements, that the costs per patient over their last years of life are 26,000 euros, for a total of 13.5 million euros.

One of the most important aspects of palliative care is the comfort of the patients as well as their feelings in the care.

In order to best meet the expectations of cancer patients, some offer early palliative care that is effective in improving both the quality of life of the patient and its life expectancy.

Osteopathy is a manual alternative medicine whose goal is to restore the lack of mobility of tissues. It can be used as a complementary treatment when a specific support is put in place. The purpose of this study is to examine the effectiveness of osteopathy in the reduction of pain in adult patients in palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (age> 18) male or female
* Patient hospitalized or admitted to a day hospital that can be followed
* EVA between 40/100 and 60/100
* Signed informed consent

Exclusion Criteria:

* Patients requiring a modification of analgesic molecule during the study.
* Clinical stability of the patient estimated during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analog Scale) evaluation (0 to 100) | day 6
  Evolution of the score of the Visual Analogue Scale (VAAS) on 100 between D0 and D6 and D0 and D1, D0 and D2, D0 and D3, D0 and D4, D0 and D5

SECONDARY OUTCOMES:
Dose of analgesic (g) | day 6
  Variation of the analgesic intake between D0 and D6 and D0 and D1, J1 and D2, J2 and D3, D3 and D4, D4 and D5, D5 and D6.
QLQ (Quality of life questionnaire) C15 Pal score | days 6
  Variation of the quality of life questionnaire (QLQ) C15 Pal score between D0 and D6

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No